CLINICAL TRIAL: NCT01509300
Title: HLA-haploidentical Allogeneic Hematopoietic Cell Transplantation Using CD3 Depletion for Children and Adolescents With Acute Leukemia, Myelodysplastic Syndrome and Solid Tumors After Conditioning of TBI, Fludarabine, Cyclophosphamide and Antithymocyte Globulin
Brief Title: HLA-haploidentical Hematopoietic Stem Cell Transplantation for Children and Adolescents With Acute Leukemia, Myelodysplastic Syndrome and Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ho Joon Im, Principal investigator, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMCPHO-SCT0902
Record Dates: First submitted 2012-01-05; First posted 2012-01-13 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Acute Leukemia; Myelodysplastic Syndrome; Solid Tumors
Keywords: TBI; Fludarabine; CD3 depletion; Children and adolescents; Haploidentical hematopoietic stem cell transplantation
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Antilymphocyte Serum; Filgrastim; Whole-Body Irradiation; fludarabine; Cyclophosphamide; Tacrolimus; Mycophenolic Acid; Rituximab

ARMS (1):
- HAPLO (Experimental)
  Interventions: Biological: anti-thymocyte globulin; Biological: filgrastim; Radiation: Total body irradiation; Drug: Fludarabine; Drug: cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Drug: Rituximab

INTERVENTIONS:
Biological: anti-thymocyte globulin — On days -10 to -9
Biological: filgrastim — Beginning on day 4 and continuing until blood counts recover
Radiation: Total body irradiation — 2Gy D-6 to D-4
Drug: Fludarabine — 30mg/M2 once daily IV on days -8 to -4
Drug: cyclophosphamide — 60 mg/kg IV on day-3 and -2
Drug: Tacrolimus — begin on 0
Drug: Mycophenolate mofetil — begin on 0
Drug: Rituximab — 375mg/m2 on day +21

SUMMARY:
RATIONALE: Conditioning with total body irradiation (TBI) and fludarabine, cyclophosphamide and anti-thymocyte globulin may induce the engraftment cross the immunologic barrier in the setting of HLA-haploidentical allogeneic hematopoietic cell transplantation. In addition, T-cell depletion may contribute to prevent developing severe acute graft versus host disease (GVHD) in haploidentical transplantation.

PURPOSE: This phase I/II trial is to evaluate the safety and efficacy of TBI, fludarabine, cyclophosphamide and antithymocyte globulin with T-cell depleted graft from haploidentical donors in treating patients with acute leukemia and myelodysplastic syndrome.

ELIGIBILITY:
Inclusion Criteria

1. Disease characteristics

   * Acute lymphoblastic leukemia (first remission, high risk; beyond first remission; refractory)
   * Acute myeloblastic leukemia (first remission, high risk; beyond first remission; refractory)
   * Myelodysplastic syndrome
   * Solid tumors (Refractory/relapse)
2. No HLA-identical family member or closely matched (8 or 7 of 8 HLA-locus match) unrelated marrow donor available
3. HLA-haploidentical related donor available

Exclusion criteria

1. Active fungal infections
2. HIV positive
3. Pregnant or nursing

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Transplantation-related mortality and overall survival of TBI, Fludarabine, Cyclophosphamide and anti-thymocyte globulin for engraftment of CD3 depleted haploidentical peripheral blood stem cells. | 2 years post-transplant

SECONDARY OUTCOMES:
Engraftment and graft failure rates | 28 days engraftment and graft failure
  Number of patients who failed to stable engraftment by 28 days
Incidence of acute GVHD | 100 days post-transplant
  Number of patients with acute GVHD.
Treatment related mortality | 100 days post-transplant
  Number of death after transplantation
Relapse rate and overall survival | 2 year after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Ho Joon Im, MD & PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Koh KN, Im HJ, Kim BE, Choi ES, Jang S, Kwon SW, Park CJ, Seo JJ. Haploidentical haematopoietic stem cell transplantation using CD3 or CD3/CD19 depletion and conditioning with fludarabine, cyclophosphamide and antithymocyte globulin for acquired severe aplastic anaemia. Br J Haematol. 2012 Apr;157(1):139-42. doi: 10.1111/j.1365-2141.2011.08924.x. Epub 2011 Nov 5. No abstract available. PMID 22055111
- [Background] Lang P, Handgretinger R. Haploidentical SCT in children: an update and future perspectives. Bone Marrow Transplant. 2008 Oct;42 Suppl 2:S54-9. doi: 10.1038/bmt.2008.285. PMID 18978746
- [Derived] Im HJ, Koh KN, Suh JK, Lee SW, Choi ES, Jang S, Kwon SW, Park CJ, Seo JJ. Refinement of treatment strategies in ex vivo T-cell-depleted haploidentical SCT for pediatric patients. Bone Marrow Transplant. 2015 Feb;50(2):225-31. doi: 10.1038/bmt.2014.232. Epub 2014 Oct 13. PMID 25310303